CLINICAL TRIAL: NCT02326207
Title: Weekly Versus no Routine Ventilator Circuit Changes in Neonatal Intensive Care Unit: Prospective, Randomized Study
Brief Title: Weekly Versus no Routine Ventilator Circuit Changes in NICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: very low enrolled participants
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Anucha Thatrimontrichai, Mr, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PSU 2014
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: Infant, Newborn; Neonatal intensive care unit; Ventilator circuit
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weekly ventilator circuit change (Experimental): Ventilator circuit change every 7 days until extubation
  Interventions: Device: Infant Ventilator Circuit Dual Heated with Autofeed Chamber
- No routine ventilator circuit change (Active Comparator): No routine ventilator circuit change until soiling or malfunction or extubation
  Interventions: Device: Infant Ventilator Circuit Dual Heated with Autofeed Chamber

INTERVENTIONS:
Device: Infant Ventilator Circuit Dual Heated with Autofeed Chamber
  Other Names: Evaqua2, RT265

SUMMARY:
The purpose of this study is to determine incidence of ventilator-associated pneumonia compared between weekly and no routine ventilator circuit changes in neonatal intensive care unit

DETAILED DESCRIPTION:
Parents were received informed consent. Enrolled neonates was randomly assigned to 2 groups as 7-day ventilator circuit change and no change group by computerization with allocated of concealment. The investigation team opened the next sequentially numbered study pack, which was stored in the neonatal unit. The assignment sequence was generated with balance within random block sizes of 4. Stratification according to birthweight was done before randomization to control for differences in patient populations. Patient characteristics were recorded as gestational age, sex, birthweight, underlying disease, date of intubation, date of extubation, duration of mechanical ventilator, reintubation, length of hospital stay, parenteral nutrition, medication (H2-blocker, PPI, narcotic drugs), transfusion and oral immune therapy. Laboratory data and radiographic data were recorded. Both groups received similarly care as the nurse was assigned to take care of patient in ratio 1-2 patients: 1 nurse, new disposable circuits were use in both groups and the VAP prevention protocol and the endotracheal suctioning protocol which followed by an American Academy of Respiratory Care (AARC) clinical practice guidelines were performed in both groups.

When the VAP was suspected the radiographic data were reviewed by two pediatric radiologists on the day of diagnosis, 3 days prior to the diagnosis and/or 2 and 7 days after diagnosis to confirm diagnosis of VAP if there is different in the results, the consensus must be made.

ELIGIBILITY:
Inclusion Criteria:

* All neonates who admitted at neonatal intensive care unit (NICU) and required ventilator support with both intubated at time of neonatal resuscitation and within the NICU as indicated

Exclusion Criteria:

* Patient was extubated or died within 2 calendar days of endotracheal intubation
* Pneumonia was diagnosed before intubation
* Outborn who was intubated before referred
* Parents declined to participate
* Incompatibility of disposable circuits and ventilator
* Chromosome abnormality or moribund

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
incidence of ventilator-associated pneumonia (percentage of ventilator-associated pneumonia (events)/mechanically ventilated infant) | within the first 30 days (plus or minus 7 days) after extubation
  percentage of ventilator-associated pneumonia (events)/mechanically ventilated infant

SECONDARY OUTCOMES:
incidence of ventilator-associated pneumonia (ventilator-associated pneumonia (events)/1,000 ventilator days) | within the first 30 days (plus or minus 7 days) after extubation
  ventilator-associated pneumonia (events)/1,000 ventilator days
Mortality rate | within the first 30 days (plus or minus 7 days) after discharge
  pneumonia-specific mortality within 7 days and at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Anucha Thatrimontrichai, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Background] Cernada M, Aguar M, Brugada M, Gutierrez A, Lopez JL, Castell M, Vento M. Ventilator-associated pneumonia in newborn infants diagnosed with an invasive bronchoalveolar lavage technique: a prospective observational study. Pediatr Crit Care Med. 2013 Jan;14(1):55-61. doi: 10.1097/PCC.0b013e318253ca31. PMID 22791095
- [Background] Apisarnthanarak A, Holzmann-Pazgal G, Hamvas A, Olsen MA, Fraser VJ. Ventilator-associated pneumonia in extremely preterm neonates in a neonatal intensive care unit: characteristics, risk factors, and outcomes. Pediatrics. 2003 Dec;112(6 Pt 1):1283-9. doi: 10.1542/peds.112.6.1283. PMID 14654598
- [Background] Afjeh SA, Sabzehei MK, Karimi A, Shiva F, Shamshiri AR. Surveillance of ventilator-associated pneumonia in a neonatal intensive care unit: characteristics, risk factors, and outcome. Arch Iran Med. 2012 Sep;15(9):567-71. PMID 22924377
- [Background] Kawanishi F, Yoshinaga M, Morita M, Shibata Y, Yamada T, Ooi Y, Ukimura A. Risk factors for ventilator-associated pneumonia in neonatal intensive care unit patients. J Infect Chemother. 2014 Oct;20(10):627-30. doi: 10.1016/j.jiac.2014.06.006. Epub 2014 Jul 4. PMID 25000829
- [Background] Han J, Liu Y. Effect of ventilator circuit changes on ventilator-associated pneumonia: a systematic review and meta-analysis. Respir Care. 2010 Apr;55(4):467-74. PMID 20406515
- [Background] Makhoul IR, Kassis I, Berant M, Hashman N, Revach M, Sujov P. Frequency of change of ventilator circuit in premature infants: Impact on ventilator-associated pneumonia. Pediatr Crit Care Med. 2001 Apr;2(2):127-132. doi: 10.1097/00130478-200104000-00006. PMID 12797871